CLINICAL TRIAL: NCT06813040
Title: Efficacy of Repetitive Transcranial Magnetic Stimulation in Chronic Pain in Patients with Temporomandibular Disorders.
Brief Title: Efficacy of Repetitive Transcranial Magnetic Stimulation in Temporomandibular Disorders.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Miguel Castelo-Branco, Full Professor, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ICNAS-FM-10,2022
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Temporomandibular Joint Disorders; TMJ disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active rTMS (Active Comparator): Repetitive transcranial magnetic stimulation over motor cortex.
  Interventions: Device: Active rTMS
- Sham rTMS (Sham Comparator): Sham repetitive transcranial magnetic stimulation over motor cortex.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS — Repetitive TMS will be applied at 10Hz on the motor cortex. The protocol consists of 2000 pulses per session and an intensity of 90% of the resting motor threshold. There will be 10 sessions with a minimum interval of 24 hours and a maximum of 72 hours. A figure-8 coil will be used.
  Arms: Active rTMS
Device: Sham rTMS — The sham TMS will have the same visual and sound characteristics, but without the passage of the magnetic field to the scalp.
  Arms: Sham rTMS

SUMMARY:
Temporomandibular disorder (TMD) refers to a group of musculoskeletal conditions that affect the temporomandibular joint (TMJ), the masticatory muscles, and the associated structures. It is assumed that 30 to 40% of cases of acute painful TMD becomes chronic. Chronic pain is a significant public health problem, affecting professional and social activities, emotional state, and quality of life. The pathophysiological mechanisms involved in chronic orofacial pain are complex and multifaceted and not yet fully understood. The coexistence of psychological factors associated with vast peripheral and central mechanisms makes chronic orofacial pain treatment a complex challenge. Due to the complexity of chronic TMDs, some patients remain refractory to current therapeutic methods. Thus, several efforts have been made to develop therapies aimed at the treatment of neuroplastic changes induced by chronic pain. In this sense, transcranial stimulation methods appear to be a promising technique. Transcranial Magnetic Stimulation (TMS) is a non-invasive, safe, and approved treatment for clinical use in psychiatric disorders such as depression and chronic pain. Given the above, it is necessary to develop studies to investigate the TMS effectiveness in chronic TMD. This study aims to evaluate the effectiveness of transcranial magnetic stimulation in patients with chronic temporomandibular disorders. An additional objective is to determine possible predictors for treatment success based on the assessment of functional brain connectivity and psychosocial characteristics.

DETAILED DESCRIPTION:
Temporomandibular disorder (TMD) is a generic term used to describe musculoskeletal disorders that affect the temporomandibular joint (TMJ), masticatory muscles, and related structures. TMD comprises two main groups: intra-articular TMD and masticatory muscle disorders. It is noteworthy that each of these groups still contains different diagnoses. Furthermore, masticatory muscle disorders and intra-articular TMD often coexist in the same individual. Such characteristics contribute to the complex diagnosis and treatment of TMDs.

It is estimated that TMD affects 5 to 12% of the population and is considered the second most prevalent musculoskeletal disorder, behind only chronic low back pain. Pain, joint noises, and limitation of mandibular movements are the main signs and symptoms of TMD. TMJ noises and limited jaw movements are often associated with intra-articular TMD. On the other hand, pain is a common symptom in different types of TMD, and it can be localized or diffuse and even as otalgia or headache. It is assumed that 30 to 40% of cases of acute painful TMD becomes chronic. Chronic pain impacts professional and social activities, emotional state, and quality of life. The pathophysiological mechanisms of chronic orofacial pain are complex and multifaceted, and not yet fully understood. In addition, the coexistence of psychological factors associated with the vast number of peripheral and central mechanisms (for example, functional and structural neuroplasticity and, more specifically, peripheral and central sensitization) makes the treatment of chronic orofacial pain a challenge extremely complex.

TMD treatment comprises a wide range of therapeutic modalities. Conservative treatments constitute the first therapeutic option, aiming to reduce joint and muscle overload, control local inflammatory factors, and reduce some risk factors, such as waking bruxism and psychological disorders. However, due to the complexity of chronic TMDs, some patients remain refractory to current therapeutic methods. Thus, several efforts have been made to develop therapies to treat neuroplastic changes associated with chronic pain. In this regard, transcranial stimulation methods appear to be a promising treatment. Transcranial Magnetic Stimulation (TMS) is a non-invasive, safe, and approved method for clinical use in psychiatric disorders and chronic pain. Recent scientific evidence has demonstrated that high-frequency TMS when applied to the motor cortex (M1), presents short-term effectiveness in reducing chronic pain and improving quality of life. A systematic review conducted by Ferreira demonstrated promising results of TMS in orofacial pain.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes, literate, aged over 18 years with the diagnosis of muscular and/or joint TMD by the Diagnostic Criteria for Temporomandibular Disorders (DC-TMD).
* Pain duration longer than 6 months.
* Intensity of orofacial pain greater than 5 on the visual analogue scale (VAS).

Exclusion Criteria:

* Volunteers who present verbal communication impairment due to a neurological disorder, a sequel to a previous illness, or a psychiatric condition.
* Pregnant women
* Individuals with any impediment to MRI: having a pacemaker or implantable defibrillator, cochlear implant, ferromagnetic aneurysm clips, electrodes used for deep brain stimulation, ocular implants, Swan-Ganz catheter, orthopedic prostheses or metallic bodies close to the area of interest.
* Individuals with any contraindication for transcranial magnetic stimulation: have focal or generalized encephalopathies, increased intracranial pressure, and severe heart disease; history of head trauma, epilepsy, and individuals with first-degree relatives diagnosed with idiopathic epilepsy; use of drugs that lower the seizure threshold (tricyclic antidepressants and antipsychotics); chronic use of alcohol or epileptogenic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Primary outcomes will be assessed before and after all TMS sessions. Follow-up will be carried out one week, two weeks, and 1 month after treatment.
  Visual Analogue Scale Visual Analogue Scale ranges from 0 to 10 and consists of a 100 mm horizontal line. The left end is labeled 'No pain,' while the right end is marked 'Worst pain imaginable
Functional limitation | Primary outcomes will be assessed before and after all TMS sessions. Follow-up will be carried out one week, two weeks, and 1 month after treatment.
  Visual Analogue Scale The Visual Analogue Scale (VAS) ranges from 0 to 10 and consists of a 100 mm horizontal line. The left end is labeled 'No functional limitation,' while the right end is marked 'Worst functional limitation imaginable.

SECONDARY OUTCOMES:
Disability associated with pain | Change from baseline to mid-treatment, immediately after the last simulated or active TMS session, and follow-up will be carried out one week, 15 days and 1 month after the end of treatment.
  Graded Chronic Pain Scale version 2.0
Depression | Change from baseline to mid-treatment, immediately after the last simulated or active TMS session, and follow-up will be carried out one week, 15 days and 1 month after the end of treatment.
  Patient Health Questionnaire - PQ-9;
Anxiety | Change from baseline to mid-treatment, immediately after the last simulated or active TMS session, and follow-up will be carried out one week, 15 days and 1 month after the end of treatment.
  Generalized Anxiety Disorder 7 - GAD-7
Central sensitization | hange from baseline to mid-treatment, immediately after the last simulated or active TMS session, and follow-up will be carried out one week, 15 days and 1 month after the end of treatment.
  Central Sensitization Inventory
Quality of Life | Change from baseline to mid-treatment, immediately after the last simulated or active TMS session, and follow-up will be carried out one week, 15 days and 1 month after the end of treatment.
  World Health Organization Quality of Life Assessment Tool - WHOQOL The WHOQOL-BREF instrument assesses the quality of life across four domains: physical, psychological, social relationships, and environment. The questionnaire provides a score for each domain, as well as an overall score derived from all domains. All scores follow a positive, increasing order, with higher scores indicating a better quality of life.
Functional connectivity | Change from baseline to one week after the end of treatment.
  Functional magnetic resonance imaging (fMRI)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Castel-Branco, PhD, Study Director — ICNAS - Institute of Nuclear Sciences Applied to Health; Catarina Duarte, PhD, Principal Investigator — ICNAS - Institute of Nuclear Sciences Applied to Health; Natália Ferreira, PhD, Principal Investigator — University of Coimbra
Locations (1):
- University of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okeson JP, de Leeuw R. Differential diagnosis of temporomandibular disorders and other orofacial pain disorders. Dent Clin North Am. 2011 Jan;55(1):105-20. doi: 10.1016/j.cden.2010.08.007. PMID 21094721
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Lovgren A, Haggman-Henrikson B, Visscher CM, Lobbezoo F, Marklund S, Wanman A. Temporomandibular pain and jaw dysfunction at different ages covering the lifespan--A population based study. Eur J Pain. 2016 Apr;20(4):532-40. doi: 10.1002/ejp.755. Epub 2015 Aug 27. PMID 26311138
- [Background] Rammelsberg P, LeResche L, Dworkin S, Mancl L. Longitudinal outcome of temporomandibular disorders: a 5-year epidemiologic study of muscle disorders defined by research diagnostic criteria for temporomandibular disorders. J Orofac Pain. 2003 Winter;17(1):9-20. PMID 12756926
- [Background] Cohen SP, Mao J. Neuropathic pain: mechanisms and their clinical implications. BMJ. 2014 Feb 5;348:f7656. doi: 10.1136/bmj.f7656. PMID 24500412
- [Background] Yin Y, He S, Xu J, You W, Li Q, Long J, Luo L, Kemp GJ, Sweeney JA, Li F, Chen S, Gong Q. The neuro-pathophysiology of temporomandibular disorders-related pain: a systematic review of structural and functional MRI studies. J Headache Pain. 2020 Jun 19;21(1):78. doi: 10.1186/s10194-020-01131-4. PMID 32560622
- [Background] de Souza RF, Lovato da Silva CH, Nasser M, Fedorowicz Z, Al-Muharraqi MA. Interventions for the management of temporomandibular joint osteoarthritis. Cochrane Database Syst Rev. 2012 Apr 18;2012(4):CD007261. doi: 10.1002/14651858.CD007261.pub2. PMID 22513948
- [Background] Greene CS, Manfredini D. Transitioning to chronic temporomandibular disorder pain: A combination of patient vulnerabilities and iatrogenesis. J Oral Rehabil. 2021 Sep;48(9):1077-1088. doi: 10.1111/joor.13180. Epub 2021 Jun 3. PMID 33966303
- [Background] O'Connell NE, Marston L, Spencer S, DeSouza LH, Wand BM. Non-invasive brain stimulation techniques for chronic pain. Cochrane Database Syst Rev. 2018 Mar 16;3(3):CD008208. doi: 10.1002/14651858.CD008208.pub4. PMID 29547226
- [Background] Ferreira NR, Junqueira YN, Correa NB, Fonseca EO, Brito NBM, Menezes TA, Magini M, Fidalgo TKS, Ferreira DMTP, de Lima RL, Carvalho AC, DosSantos MF. The efficacy of transcranial direct current stimulation and transcranial magnetic stimulation for chronic orofacial pain: A systematic review. PLoS One. 2019 Aug 15;14(8):e0221110. doi: 10.1371/journal.pone.0221110. eCollection 2019. PMID 31415654